CLINICAL TRIAL: NCT05085457
Title: The Use of ExPreS - Extubation Predictive Score - in the Weaning of Patients in Invasive Mechanical Ventilation: a Randomized Clinical Trial
Brief Title: The Use of ExPreS in the Weaning of Patients in Invasive Mechanical Ventilation
Acronym: ExPreS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Oeste de Santa Catarina (Other)
Responsible Party: Principal Investigator, Antuani Rafael Baptistella, Professor, Universidade do Oeste de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: RCT ExPreS
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Insufficiency
Keywords: Mechanical Ventilation; Extubation; Weaning
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive the intervation of Control group or ExPreS group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant will not know if the ExPreS or just RSBI were calculated before extubation. The SBT will be the same for both groups.
  Investigator and outcomes assessor will not have access to whole patients' data, just the primary and secundary outcomes to perform the statistical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): On group I (T-ayre and standard protocol), SBT must begin with the pacient in T-ayre, oxygen support that is proprotional to the fraction of inspired oxygen in invasive mechanical ventilation (IMV), during 30 minutes. If the pacient does not show any sign of SBT failure, the rapid shallow beathing index (RSBI) will be calculated and pacients with RSBI lower than 105 L/min will be extubated, meanwhile pacients with RSBI higher than 105 L/min will return to MV for at least 24 hours until the perfomance of a new SBT.
- ExPreS Group (Experimental): On group II (T-ayre and ExPreS protocol), the pacient will be submitted to the SBT with T-ayre, with oxygen support that is proprotional to the fraction of inspired oxygen in IMV, during 30 minutes. If the pacient does not show any sign of SBT failure, ExPreS will be calculated. If punctuation is lower than or equal to 44, it indicates weaning failure and the pacient mjust return to MV for 24 hours at least. Punctuation between 45 and 58 must be evaluated if the pacient presents chronic obstructive pulmonary desease (COPD), obesity or heart desease. In this case, the weaning must be continued if there isn't any risck factors. Punctuation higher than or equal 59 indicates that the pacient can be extubated.
  Interventions: Diagnostic Test: ExPreS Protocol

INTERVENTIONS:
Diagnostic Test: ExPreS Protocol — the pacient will be submitted to the SBT with T-ayre, with oxygen support that is proprotional to the fraction of inspired oxygen in IMV, during 30 minutes. If the pacient does not show any sign of SBT failure, ExPreS will be calculated. If punctuation is lower than or equal to 44, it indicates weaning failure and the pacient mjust return to MV for 24 hours at least. Punctuation between 45 and 58 must be evaluated if the pacient presents chronic obstructive pulmonary desease (COPD), obesity or heart desease. In this case, the weaning must be continued if there isn't any risck factors. Punctuation higher than or equal 59 indicates that the pacient can be extubated.
  Arms: ExPreS Group

SUMMARY:
Patients on mechanical ventilation (MV) must undergo weaning, an interruption of ventilatory support. Several scores have been developed to predict this outcome, but the failure index in weaning and extubation remains high. The aim of this study is to evaluate the effect of ExPreS - Extubation Predictive Score - on the rate of successful extubation. This research will be conducted in a randomized clinical trial in ICUs of several hospitals. It is expected that there will be a difference between devices for predicting extubation success, and because ExPreS is a protocol that evaluates various parameters related to many organs and systems, it has a better ability to predict extubation success in MV patients.

DETAILED DESCRIPTION:
1. OBJECTIVES

1. 1 General To evaluate the effect of the Extubation Predictive Score (ExPreS) on the rate of successful extubation.

   1.2 Specific To compare the predictive ability of ExPreS with the standard protocol at the study site.

   To determine the success and failure rate of extubation within 48 hours according to the protocols used.
2. SELECTION OF PARTICIPANTS The sample will be composed of patients admitted to the ICUs of the participating institutions, on MV for more than 24 hours. Inclusion criteria are pacients admitted to the ICU, older than 18 years and on MV for more than 24 hours. The free and informed consent form must be signed by a family member or responsible adult. Exclusion criteria are death before SBT, tracheostomy, self-extubation, accidental extubation and failure to sign the consent form. The patient who fails extubation and requires reintubation will not be randomized.
3. RANDOMIZATION Patients meeting the criteria for initiation of MV weaning - improvement of the condition causing respiratory failure; arterial oxygen partial pressure higher than 60 mmHg, with inspired oxygen fraction lower than 0. 4 and positive end-expiratory pressure of 5 cm of water or less; hemodynamically stable (no or low dose of vasopressors, absence of decompensated coronary insufficiency or arrhythmias with hemodynamic repercussions); patient's ability to initiate an inspiratory effort; Absence of significant acid-base imbalance, tolerating PSV mode with PEEP of 3-5 and pressure over the PEEP of 7 cmH2O with adequate ventilation (volume of 6 ml/kg and RR ˃ 35/min) - will meet the conditions and will be randomized and submitted to SBT.

   Randomization will be performed using the program www.random.org and, for allocation concealment The numbers generated will be placed in sealed and opaque envelopes with the previously defined nomenclature for each group: Group I (T-ayre and standard protocol) and Group II (T-ayre and ExPreS protocol). The envelopes are numbered and placed in order. Therefore, the evaluator and the researchers are prevented from choosing the group to which the individual will be assigned. Only one person will be responsible for opening the envelope and informing the witch group to which he or she has been assigned.
4. INTERVENTION Patients will be assigned to different interventions according to each group. Failure criteria for SBT will be the same for all groups: agitation, anxiety, decreased level of consciousness, respiratory rate higher than 35/min and/or use of accessory muscles, oxygen saturation measured by pulse oxymetry lower than 90% with fraction of inspired oxygen lower than 0.4 more than 0.5, heart rate higher than 140 bpm or an increase higher than 20% of basal, systolic blood pressure (SBP) lower than 90 mmHg or higher than 180 mmHg or presenting arrhythmia after initiation of SBT.

   In group I (T-Aire and standard protocol), SBT must begin with the patient in T-Aire, oxygen support proportional to the fraction of inspired oxygen during invasive mechanical ventilation (IMV), for 30 minutes. If the patient shows no signs of SBT failure, the rapid shallow breathing index (RSBI) is calculated and patients with RSBI less than 105 L/min are extubated, while patients with RSBI greater than 105 L/min are returned to MV for at least 24 hours until a new SBT is performed.

   In group II (T-ayre and ExPreS protocol), the patient is subjected to SBT with T-ayre with oxygen support proportional to the fraction of inspired oxygen in IMV for 30 minutes. If the patient shows no signs of SBT failure, ExPreS is calculated. A punctuation less than or equal to 44 indicates weaning failure and the patient must return to MV for at least 24 hours. Punctuation between 45 and 58 must be evaluated if the patient has chronic obstructive pulmonary disease (COPD), obesity, or heart disease. In this case, weaning must be continued if there are no risk factors. A score greater than or equal to 59 indicates that the patient can be extubated.

   Patients in both groups are assessed for airway patency using the cuff leak test. Patients with a difference of more than 10% between inspiratory and expiratory tidal volumes can be extubated.
5. OUTCOME The primary outcome in both groups is successful extubation at 48 hours. To be considered positive, the patient must remain without the need to return to MV for at least 48 hours and must not require NIV for the next 48 hours after extubation. Secondary outcomes are reintubation, ICU length of stay, hospital length of stay, and in-hospital mortality.
6. RESEARCH INSTRUMENTS The instruments for data collection are forms designed by the researchers. The choice of the form will be made by randomization, which will take place after 24 hours of MV with endotracheal tube, according to the inclusion and exclusion criteria.
7. DATA ANALYSIS Collected data will be tabulated on Microsoft Excel program and statistical analysis will be made on IBM SPSS statistics, v25 and GraphPad Prism 6 programs.
8. ETHICAL ASPECTS This project has been submitted to the Research Commission of the Hospital Institution of Interest for authorization to conduct the research and to the Research Ethics Committee of Unoesc, and it has been approved by number 4.524.592 (CAAE 39925920.0.0000.5367). It will follow the ethical principles of the resolution number 466/2021, of the Nacional Health Council. The research will have commitment with data privacy and confidentiality, by preserving the anonymity of the participants.

This research is classified as low risk for the research participants, causing little discomfort to the patient, which is justified by the expected benefit. There will be no intervention or intentional modification of physiological or psychological and social variables of individuals who participate in the study.

The benefits of participation are indirect for the patients, although by demonstrating a better outcome, the study proposes a better testing of protocols that will contribute to the elaboration of strategies to achieve a better extubation success.

The consent to participate in the study will be formalized by signing the free and informed consent form, which will be given in two copies, one for the family member or responsible person and one for the researchers, according to Resolution 466/2021, of the Nacional Health Council.

In order to maintain the safety of all individuals, precautionary measures will be adopted for the transmission of COVID-19. Hands will be disinfected with 70% alcohol when entering the institution, before and after entering the ICU and before manipulating documents. Masks will be used at all times.

ELIGIBILITY:
Inclusion Criteria:

* Pacients admitted in ICU that are more than 18 years;
* MV for more than 24 hours;
* Assignature of the free and informed consent form by a family member or responsable adult.

Exclusion Criteria:

* Death before SBT;
* Tracheostomy;
* Self-extubation;
* Accidental extubation;
* Absence of signature of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Extubation Success | 48 hours
  No reintubation nor dependence of NIV

SECONDARY OUTCOMES:
Reintubation | 28 days
  Need of reintubation
IMV lenght of stay | 28 days
  Time in need of IMV
ICU lenght of stay | 28 days
  Time in need of ICU
Hospital lenght of stay | 28 days
  Time in hospital stay
In Hospital mortality | 28 days
  Outcome in hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário Santa Terezinha, Joaçaba, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No